CLINICAL TRIAL: NCT00777816
Title: A Blinded, Placebo-controlled, Study of the Safety and Pharmacokinetics of XOMA 052 Administered to Subjects With Active, Stable, Moderate to Severe Rheumatoid Arthritis
Brief Title: Safety and Pharmacokinetics Study of XOMA 052 in Subjects With Active, Stable, Moderate to Severe Rheumatoid Arthritis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Alan M. Solinger, M.D. / Medical Monitor; V.P. Clinical Immunology, XOMA (US) LLC
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: X052070
Record Dates: First submitted 2008-10-17; First posted 2008-10-22 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: XOMA 052
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XOMA 052 — A single dose of study drug on Day 0, administered either as an intravenous (IV) infusion or as a subcutaneous (SC) injection.
  Arms: 1
Drug: Placebo — A single dose of placebo on Day 0, administered either as an intravenous (IV) infusion or as a subcutaneous (SC) injection.
  Arms: 2

SUMMARY:
Study X052070 will evaluate the safety and pharmacokinetics (PK) of XOMA 052 administered to patients with active, stable, moderate to severe rheumatoid arthritis (RA).

It is hypothesized that administration of XOMA 052 is likely to improve inflammatory control in subjects with RA.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology (ACR) diagnostic criteria for RA
* Moderate to severe disease, defined as follows - At least six tender and six swollen joints (28 joint count) AND ESR > 28 mm/hr or CRP > 1.0 mg/dL
* Current duration of RA at Screening ≥ 6 months and ≤ 20 years
* RA and other medical conditions must be stable.
* Age ≥ 18 and ≤ 75 at Screening
* Weight ≥ 80 lbs (36.3 kg) and ≤ 275 lbs (125.0 kg)
* For females with child-bearing potential, a negative serum pregnancy test

Exclusion Criteria:

* Major surgery within 28 days prior to Day 0
* Joint replacement surgery within 60 days prior to Day 0 or joint replacement surgery planned within 9 months following Day 0
* Known HIV antibody, or hepatitis B surface antigen
* History of malignancy within 5 years prior to Screening other than carcinoma in situ of the cervix, or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin
* Immunodeficiency
* History or symptoms of a demyelinating disease
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies. Respiratory distress (dyspnea, oxygen desaturation with pO2 < 90% or onset of acute respiratory distress syndrome), flank or back pain, and/or hypotension may be signs of anaphylaxis.
* History of tuberculosis, positive PPD test, active atopic disease requiring medication, or asthma. A subject who has had a positive PPD test but has completed a course of treatment for tuberculosis, had a documented vaccination against tuberculosis, or had a negative QuantiFERON -TB test result is eligible.
* Chronic obstructive pulmonary disease (COPD), asthma, or other pulmonary disease requiring more therapy than using one inhaler 4× daily
* Significant systemic involvement secondary to RA (e.g. vasculitis, pulmonary fibrosis)
* Liver disease (e.g., hepatitis, cirrhosis) or abnormal hepatic function. If the diagnosis of liver disease was based on positive Hep C serology due to prior vaccination, the subject is eligible.
* Pregnant or planning to become pregnant during the course of the study, or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-02; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety assessed by pre- and post-treatment serial measurements of vital signs, clinical laboratory assessments, and treatment-emergent adverse events. | Day 0 pre-dose through Day 56

SECONDARY OUTCOMES:
Pharmacokinetic assessments from serum samples collected at time points specified in the protocol. | Day 0 Pre-dose through Day 56
Assessment of inflammatory markers CRP and ESR collected at time points specified in the protocol. | Day 0 pre-dose through Day 56
Assessment of Rheumatoid Arthritis disease status by the collection of ACR (American College of Rheumatology) core criteria at time points specified in the protocol. | Day 0 pre-dose through Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Alan Solinger, M.D., Study Director — XOMA (US) LLC
Locations (2):
- United States (2):
  - Clearwater, Florida
  - Middleburg Heights, Ohio